CLINICAL TRIAL: NCT06017245
Title: Could the Bone-Myoregulation Reflex Explain the Development of Sarcopenia in Postmenopausal and Senile Osteoporosis?
Brief Title: The Bone-Myoregulation Reflex and Development of Sarcopenia in Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BMROPS
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Sarcopenia; Osteoporosis
Keywords: muscle strength; bone mineral density
MeSH Terms: conditions — Sarcopenia; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Healthy young-adult groups
  Interventions: Device: whole-body vibration to Control
- Senile osteoporosis (Experimental): Patients with senile osteoporosis
  Interventions: Device: whole-body vibration to Control
- Postmenopausal osteoporosis (Experimental): Patients with postmenopausal osteoporosis
  Interventions: Device: whole-body vibration to Control

INTERVENTIONS:
Device: whole-body vibration to Control — Whole-body vibration (WBV) will be applied while standing upright. During this position, he will be asked not to voluntarily contract the calf muscles and to remain relaxed. The vibration will be applied with the PowerPlate® Pro5 WBV (London UK) device. The vibration amplitude will be 2 mm. The vibration frequency will be 30, 33, and 36 Hz. Each vibration frequency will be applied for 45 seconds. A 5-second rest period will be applied between vibrations of 45 seconds.

SUMMARY:
Bone and skeletal muscle are in a single unit that interacts with each other structurally and functionally. The aim of this study is to determine the contribution of bone myoregulation reflex as a neuronal crosstalk mechanism on the development of sarcopenia in postmenopausal and senile osteoporosis

DETAILED DESCRIPTION:
Bone and skeletal muscle are in a single unit that interacts with each other structurally and functionally. While myokines synthesized and released in skeletal muscle modulate the bone formation and destruction process, osteokines synthesized and released by bone cells have positive or negative effects on muscle (4,5,6,7,8,9). In addition to humoral crosstalk mechanisms between muscle and bone, there is also a neuronal crosstalk mechanism defined as bone myoregulation reflex. The aim of this study is to determine the contribution of bone myoregulation reflex as a neuronal crosstalk mechanism on the development of sarcopenia in postmenopausal and senile osteoporosis (10,11,12,13,14). Osteoporotic cases would be determined by standard DXA measurements.

The vibration will be applied with the PowerPlate® Pro5 whole-body vibration (London UK) device. The vibration amplitude will be 2 mm. The vibration frequency will be 30, 33, and 36 Hz. Each vibration frequency will be applied for 45 seconds. A 5-second rest period will be applied between vibrations of 45 seconds.

Surface EMG recordings will be taken from the right soleus muscle using the bipolar technique. A pair of self-adhesive Ag/AgCl (Redline®) electrodes will be adhered to the skin according to the SENIAM protocol(2). Recordings will be taken in the 1-500 Hz frequency band. Surface electromyography (EMG) recordings will be taken with a PowerLab ® (ADInstruments, Oxford, UK) data recorder with a sample rate of 20 KHz. EMG recordings will be analyzed offline with LabChart7 Pro® version 7.3.8 (ADInstruments, Oxford, UK). The acceleration measurement data will be recorded with the PowerLab (ADInstrument London) data acquisition simultaneously with the EMG recording. Acceleration recording will be made with a sample rate of 20 KHz.

ELIGIBILITY:
Inclusion Criteria:

* For healthy young adults control Healthy volunteers aged 20-45 years
* For postmenopausal osteoporosis Hip DXA T-score (neck or total hip) < -2.5
* For the Senile osteoporosis Over 65 years Male Hip DXA T-score (neck or total hip) < -2.5 Female

Exclusion Criteria:

* Osteopenic cases
* Possible sarcopenia (according to EWGSOP2 criteria)
* Vertigo
* Kidney stone
* Panic attack story
* Secondary osteoporosis
* Those with polyneuropathy, central nervous system disease clinic/history
* Myopathies (steroid, vitamin D deficiency, primary muscle diseases, etc.)
* Cases with lesions on the soleus skin
* History of fracture in lower extremity, joint prosthesis
* Lower extremity active/acute thrombophlebitis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Bone myoregulation reflex latency | up to 2 weeks
  It was defined as the period between the onset of effective mechanical stimulation and the onset of the reflex in surface electromyography.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, MD, Principal Investigator — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- Ilhan Karacan, Istanbul, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Karacan I, Cakar HI, Sebik O, Yilmaz G, Cidem M, Kara S, Turker KS. A new method to determine reflex latency induced by high rate stimulation of the nervous system. Front Hum Neurosci. 2014 Jul 18;8:536. doi: 10.3389/fnhum.2014.00536. eCollection 2014. PMID 25100978
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Karacan I, Cidem M, Cidem M, Turker KS. Whole-body vibration induces distinct reflex patterns in human soleus muscle. J Electromyogr Kinesiol. 2017 Jun;34:93-101. doi: 10.1016/j.jelekin.2017.04.007. Epub 2017 Apr 24. PMID 28457998
- [Background] Karamehmetoglu SS, Karacan I, Cidem M, Kucuk SH, Ekmekci H, Bahadir C. Effects of osteocytes on vibration-induced reflex muscle activity in postmenopausal women. Turk J Med Sci. 2014;44(4):630-8. PMID 25551934